CLINICAL TRIAL: NCT00002010
Title: Open, Non-Comparative Study of Fluconazole in Patients With Coccidioidal Meningitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 012P; 056-170
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-02

CONDITIONS: Meningitis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Fluconazole; Coccidioidin; Acquired Immunodeficiency Syndrome; Coccidioidomycosis
MeSH Terms: conditions — Meningitis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; Coccidioidomycosis | interventions — Fluconazole

INTERVENTIONS:
Drug: Fluconazole

SUMMARY:
The study is intended to examine the efficacy of fluconazole for the treatment of coccidioidal meningitis in patients with new onset of infection, relapse of previous infection, or failed previous therapy. Drug efficacy, safety and tolerance will be examined.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Immunosuppressive therapy including corticosteroids and/or cytotoxic agents.
* Antiviral therapy (e.g., zidovudine (AZT)).
* Prophylaxis for Pneumocystis carinii pneumonia (PCP).
* Any exceptions to use of concomitant medications must be approved by Pfizer Central Research prior to study entry.

Concurrent Treatment:

Allowed:

* Radiation therapy for mucocutaneous Kaposi's sarcoma.

Patients must:

* Be clinically judged to be in need of treatment for coccidioidal meningitis.
* Have > 1 week life expectancy.
* Allowed:
* Immunocompromised patients.
* Patients with renal disease will have the dose of fluconazole adjusted and serum levels may be monitored.

Prior Medication:

Allowed:

* Amphotericin B.
* Ketoconazole.
* Miconazole.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Current antifungal infection that is responding to another agent. Findings of improvement include one of the following, while on other therapy (without subsequent relapse of the item):
* CSF culture conversion from positive to negative.
* OR
* CSF antibody titer decrease of at least one dilution.
* OR
* Improvement in signs and symptoms of meningitis.
* Have received more than minimal systemic antifungal therapy (see Patient Inclusion Criteria), unless they meet criteria for previous treatment failure or relapse. They must not have received this therapy since the time relapse or failure was documented, except for minimal antifungal therapy allowed in Patient Inclusion Criteria.
* Immediately life-threatening coccidioidomycosis defined as infection of such a degree of clinical severity that the patient would be expected to die within 1 week, if untreated, based on clinical judgment.
* Experienced a prior allergic reaction or major side effect from an imidazole or triazole compound.

Concurrent Medication:

Excluded:

* Barbiturates.
* Phenytoin.
* Oral hypoglycemics.
* Coumadin type anticoagulants.
* Other systemic or intrathecal antifungal therapy.
* Other experimental agents with exceptions noted in concomitant medications section.
* Any exceptions to these prohibitions of concomitant medications must be approved by Pfizer Central Research prior to study entry.

Patients with the following are excluded:

* Are responding or are improving on current antifungal therapy with another agent.
* Have received more than minimal systemic antifungal therapy (see Patient Inclusion Criteria), unless they meet criteria for previous treatment failure or relapse. They must not have received this therapy since the time relapse or failure was documented, except for minimal antifungal therapy allowed in Patient Inclusion Criteria.
* Immediately life-threatening coccidioidomycosis defined as infection of such a degree of clinical severity that the patient would be expected to die within 1 week, if untreated, based on clinical judgment.
* Experienced a prior allergic reaction or major side effect from an imidazole or triazole compound.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Tucson Veterans Administration Med Ctr, Tucson, Arizona
  - HIV Research Group, San Diego, California
  - Audie L Murphy Veterans Administration Hosp, San Antonio, Texas